CLINICAL TRIAL: NCT02120560
Title: Uninterrupted Versus Interrupted Anticoagulation in Atrial Fibrillation Ablation - Cerebral Thromboemboli and Neurocognitive Performance
Brief Title: Anticoagulation in AF Ablation and Effects on Neurocognitive Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-13595
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation; Cerebrothromboembolus; Neurocognitive Function
Keywords: Atrial Fibrillation Ablation; Cerebrothromboemboli; Neurocognitive Function
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interrupted Anticoagulation (Active Comparator): Patients randomized to undergo atrial fibrillation ablation with interrupted anticoagulation with apixaban (5mg twice daily; 2.5mg twice daily >80 years old, Cr > 1.5, wt < 60kg), rivaroxaban (20mg daily; 15mg daily CrCl < 50 mL/minute), dabigatran (150mg twice daily; 75mg twice daily CrCl < 30mL/minute), or warfarin (dosed case-by-case).
  Interventions: Procedure: Atrial Fibrillation Ablation
- Uninterrupted anticoagulation with warfarin (Active Comparator): Patients randomized to undergo atrial fibrillation ablation with uninterrupted anticoagulation with warfarin (dosed case-by-case).
  Interventions: Procedure: Atrial Fibrillation Ablation

INTERVENTIONS:
Procedure: Atrial Fibrillation Ablation — Both treatment arms will undergo atrial fibrillation ablation.

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in the United States, and treatment by AF ablation is quickly becoming the favored definitive therapy. Nonetheless, AF ablation comes with some risk, including bleeds related to vascular access and myocardial damage, as well as the rare incidence of clinical stroke from blood clots that travel from the heart to the brain, termed "cerebrothromboemboli." In fact, cerebrothromboemboli without any symptoms have been detected by special imaging procedures called brain magnetic resonance imaging (MRI) in as many as 22% of cases.(1-6) There remains clinical equipoise amongst experts regarding balancing the risks and benefits of continued versus interrupted blood thinning, or "anticoagulation" during AF ablation as they pertain to risk of bleed and cerebrothromboemboli prevention, respectively, and the potentially more subtle sequelae of these apparently silent cerebrothromboemboli remain unknown. In fact, both interruption and continuation of anticoagulation during AF ablation are the standard of care. The investigators will perform the first randomized trial of uninterrupted versus interrupted anticoagulation in patients undergoing AF ablation to determine if it mitigates neurologic injury. The objective of this research is to investigate the effect of continued anticoagulation for AF ablation on cerebrothromboemboli, and the neurocognitive sequelae of embolic lesions, which to this point are considered subclinical. The investigators hypothesize that continued anticoagulation will both reduce cerebrothromboemboli and mitigate any potential decline in neurocognitive function post-procedurally. The investigators also hypothesize that the incidence of cerebrothromboemboli (CTE) by MRI will mediate that difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older with AF (paroxysmal or persistent) who are to undergo an elective AF ablation procedure at UCSF will be eligible for enrollment.

Exclusion Criteria:

* Patients will be excluded if they have:
* A contraindication of warfarin therapy (pregnancy, recent bleed, inability of have serial INR checks)
* A contraindication or relative contraindication to interruption of anticoagulation (e.g. mechanical valve, clotting disorder such as antiphospholipid syndrome, recent history of pulmonary embolism or history of recurrent pulmonary embolism)
* A contraindication to transesophageal echocardiogram; any contraindication to MRI
* Have a diagnosed condition of dementia or a diagnosis that precludes accurate assessment of neurocognitive function
* Non-English speakers
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke | 4 weeks
  The incidence of peri-procedural stroke will be measured.
Incidence of Cerebrothromboemboli | 1 day
  The incidence of cerebrothromboemboli post-ablation will be measured by comparing post-procedural brain MRI to pre-procedural brain MRI.
Change in Neurocognitive Performance | approximately 4 weeks
  Change in neurocognitive function will be measured by comparing performance on a battery of validated neurocognitive tests to pre-procedural performance.
Bleeding Complications | approximately 1 week
  The incidence of intra- and post-procedural bleeding complications, specifically hemopericardium and groin access complications, will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Deneke T, Shin DI, Balta O, Bunz K, Fassbender F, Mugge A, Anders H, Horlitz M, Pasler M, Karthikapallil S, Arentz T, Beyer D, Bansmann M. Postablation asymptomatic cerebral lesions: long-term follow-up using magnetic resonance imaging. Heart Rhythm. 2011 Nov;8(11):1705-11. doi: 10.1016/j.hrthm.2011.06.030. Epub 2011 Jul 2. PMID 21726519
- [Background] Gaita F, Leclercq JF, Schumacher B, Scaglione M, Toso E, Halimi F, Schade A, Froehner S, Ziegler V, Sergi D, Cesarani F, Blandino A. Incidence of silent cerebral thromboembolic lesions after atrial fibrillation ablation may change according to technology used: comparison of irrigated radiofrequency, multipolar nonirrigated catheter and cryoballoon. J Cardiovasc Electrophysiol. 2011 Sep;22(9):961-8. doi: 10.1111/j.1540-8167.2011.02050.x. Epub 2011 Mar 31. PMID 21453372
- [Background] Haeusler KG, Koch L, Herm J, Kopp UA, Heuschmann PU, Endres M, Schultheiss HP, Schirdewan A, Fiebach JB. 3 Tesla MRI-detected brain lesions after pulmonary vein isolation for atrial fibrillation: results of the MACPAF study. J Cardiovasc Electrophysiol. 2013 Jan;24(1):14-21. doi: 10.1111/j.1540-8167.2012.02420.x. Epub 2012 Aug 22. PMID 22913568
- [Background] Herrera Siklody C, Deneke T, Hocini M, Lehrmann H, Shin DI, Miyazaki S, Henschke S, Fluegel P, Schiebeling-Romer J, Bansmann PM, Bourdias T, Dousset V, Haissaguerre M, Arentz T. Incidence of asymptomatic intracranial embolic events after pulmonary vein isolation: comparison of different atrial fibrillation ablation technologies in a multicenter study. J Am Coll Cardiol. 2011 Aug 9;58(7):681-8. doi: 10.1016/j.jacc.2011.04.010. Epub 2011 Jun 12. PMID 21664090
- [Background] Ichiki H, Oketani N, Ishida S, Iriki Y, Okui H, Maenosono R, Ninomiya Y, Matsushita T, Miyata M, Hamasaki S, Tei C. Incidence of asymptomatic cerebral microthromboembolism after atrial fibrillation ablation guided by complex fractionated atrial electrogram. J Cardiovasc Electrophysiol. 2012 Jun;23(6):567-73. doi: 10.1111/j.1540-8167.2011.02259.x. Epub 2012 Feb 7. PMID 22313240